CLINICAL TRIAL: NCT04633018
Title: A Patient-Centered Asthma Management Communication Intervention for Rural Latino
Brief Title: A Patient-Centered Asthma Management Communication Intervention for Rural Latino Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Robin Dawson, Associate Professor, University of South Carolina
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1K23HL133596-01A1 (NIH)
Record Dates: First submitted 2020-11-16; First posted 2020-11-17 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Asthma
Keywords: mHealth; Latino; asthma; limited English proficiency; pediatrics; school nursing
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Patient-centered asthma intervention feasibility (Experimental): Investigate the effect of the patient-centered asthma intervention using the AsthmaMD app on school days missed and medication adherence.
  Interventions: Device: AsthmaMD mobile application
- Wait list control (Experimental): Control group with usual care (not using app).
  Interventions: Other: Usual care

INTERVENTIONS:
Device: AsthmaMD mobile application — asthma management app with Spanish-language user interface
  Arms: Patient-centered asthma intervention feasibility
Other: Usual care — Asthma management without the app
  Arms: Wait list control

SUMMARY:
The purpose of this research is to develop and evaluate an mHealth communication intervention designed to improve asthma medication adherence amongst rural Latino children in South Carolina.

DETAILED DESCRIPTION:
The overall prevalence of asthma is highest in the US south, which has one of the fastest growing Latino populations in the country. In South Carolina, asthma is the leading cause of children's hospitalization and emergency department (ED) visits, with significant direct and indirect costs. Although rates of childhood asthma are lower in Latinos (with the exception of children of Puerto Rican origin) than in whites, Latinos are more likely to have a higher incidence of uncontrolled asthma symptoms, ED visits, repeat hospitalizations, and poorer health in general. Current interventions addressing asthma control include outpatient clinic based and home visitation programs. Rural Latino families have difficulty participating with these types of programs due to work, family, and transportation constraints.

The adaptability of mobile apps holds the potential to target the unique challenges to management experienced by rural Latino children with asthma experience. The goal of this study is to develop and evaluate a patient-centered collaborative intervention between rural Latino children with asthma and their families, school-based nursing, and primary care providers, facilitated by the use of a smart phone based bilingual mobile app. The specific aims are to:

1. Produce and validate a Spanish translation of an existing asthma management app and evaluate its usability with Latino parents of children with asthma; and
2. Develop and evaluate a triadic, patient-centered asthma intervention preliminary protocol, facilitated by the bilingual mobile app validated in aim 1.

ELIGIBILITY:
Inclusion Criteria:

1) children self/family-identified as Hispanic/Latino or African American, 2) school-aged (5-18 years) and attends school within the Lancaster County School District, 3) has received a diagnosis of asthma from a health care provider and is taking a controller medication, and 4) parents/primary caregiver (e.g., grandparents, extended family) language of preference is Spanish or English.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Mobile app usability and acceptability | 1 week
  Participants with Spanish as first language use the translated app for ease of use and identification of interface problems
Preliminary protocol testing of mobile app-facilitated triadic communication | 3 months
  Develop and evaluate a triadic, patient-centered asthma intervention preliminary protocol, facilitated by the Spanish language mobile app. Post-intervention data regarding the experiences of the participants in this collaborative intervention will be obtained through a post-intervention focus group facilitated by the PI with the PCPs and school nurses, and five interviews conducted by a bilingual research assistant with the Latino families.
Investigate the feasibility of the patient-centered asthma intervention | 6 months
  Investigate the feasibility of the patient-centered asthma intervention from aim 2 using a wait list randomized control trial (RCT) to investigate the effects of the intervention on school days missed and medication adherence. Anticipated quantitative data includes the information entered into the app, encrypted, and transmitted to the school nurse by the parent/caregiver. These data will include selected NIH/AHRQ standardized asthma outcomes,47 including the primary outcome measures of medication adherence information (asthma medication ratio48 - predictive of childhood asthma ED visits and hospitalizations) and school days missed.

SECONDARY OUTCOMES:
Medication adherence and lung function tests | 6 months
  Secondary outcome measures include frequency of rescue inhaler use, as well as asthma exacerbations, outpatient clinic visits, and emergency department visits. Lung capacity will be obtained pre- and post-intervention/bronchodilation using spirometry49 to obtain relevant lung function variables such as FEV1 and FEV1/FVC. Measures from the control group will include medication counts, number of asthma exacerbations, ED/outpatient clinic visits, and spirometry measures on enrollment, during the intervention phase, and again at the end of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Robin M Dawson, PhD, Principal Investigator — University of South Carolina College of Nursing
Locations (1):
- Lancaster County School District, Lancaster, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dawson RM, Heiney SP, Messias DH, Ownby D. A Patient-Centered Asthma Management Communication Intervention for Rural Latino Children: Protocol for a Waiting-List Randomized Controlled Trial. JMIR Res Protoc. 2020 Dec 1;9(12):e18977. doi: 10.2196/18977. PMID 33258784